CLINICAL TRIAL: NCT02639208
Title: Improving Support for Older Patients Receiving Neo/Adjuvant Chemotherapy for Breast Cancer Using a Novel Social Media Intervention
Brief Title: Novel Social Media Intervention For Older Br CA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: CURE Foundation (Other)
Responsible Party: Principal Investigator, Rachel Freedman, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-326
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: Breast Cancer I; Breast Cancer Stage II; Breast Cancer Stage III
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PatientsLikeMe (PLM) (Experimental): After the screening procedures confirm eligibility.
  * Baseline Survey Assessment and PatientsLikeMe Introduction
  * Treatment Evaluation on PLM website at predetermined times per protocol
  * Final Survey
  Interventions: Other: PatientsLikeMe (PLM)

INTERVENTIONS:
Other: PatientsLikeMe (PLM)

SUMMARY:
The number of patients 60 and older with breast cancer is increasing as our population ages. Despite the fact that the majority of breast cancers occur in patients 60 and over, these patients are consistently under-represented in clinical trials. Because patients 60 and older are an under-studied group, investigators do not have detailed information on the side effects and experiences for these patients receiving chemotherapy. Understanding the side effects patients receiving chemotherapy experience is an important part of this study.

In addition, past research has shown that having poor social support can affect quality of life, mood, and outcomes for people with cancer. However, few studies in the past have focused on improving the quality of life and support systems that patients have while they receive treatment.

This research study is evaluating how engaging in an online support community may improve the experience of older patients receiving chemotherapy.

DETAILED DESCRIPTION:
This clinical trial will evaluate how an on-line health information sharing community of patients called PatientsLikeMe, www.patientslikeme.com, [or "PLM"] may help patients feel better supported during treatment. This study will also evaluate how much PLM can help collect information on side effects from chemotherapy and endocrine treatments, and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be women ≥60 years age with histologically or cytologically confirmed, stage I-III breast cancer with a treatment plan that includes any neoadjuvant or adjuvant chemotherapy(either in the context of standard treatment or a clinical trial and including chemotherapy, treatments targeting the human epidermal growth factor receptor protein 2 [HER2]), hormonal therapy or radiation.
* Enrollment must occur according to one of the following: (1) For those receiving chemotherapy/infusional therapy, patients must enroll during the 4 weeks prior to or on the day of treatment initiation, (2) For those enrolling during hormonal therapy and/or radiation, patients must enroll within 6 months of diagnosis of breast cancer, defined as the date of initial biopsy. Patient may be receiving hormonal therapy, radiation therapy, or both at the same time of enrollment, (3) Patients who did not enroll during their chemotherapy are still eligible to enroll during subsequent hormonal therapy or radiation as long as it is within 6 months of diagnosis.
* Participants must be approached before start of treatment. Patients must be able to understand, read, and write in English and be able to understand and have willingness to sign a written informed consent document.
* Patients are eligible regardless of ECOG performance status, life expectancy or, organ/marrow function.
* Patients must have the ability to access the internet at least once per week, and this can occur in the patient's home, relatives' homes, work setting, or Dana-Farber (in addition to coffee shops, libraries, etc if applicable). Having a computer is not required. An iPad will be provided to any patient who needs one for the duration of the study.

Exclusion Criteria:

* Patients with metastatic breast cancer are not eligible to participate.
* Participants who have started their treatment plan are not eligible.
* Those unable to understand, read, or write in English are not eligible.
* Men are not eligible for this study.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Feasibility/ Rate of Participant Login - PLM | 4-6 months
  We will describe the degree of patient use of the PLM platforms and the associations of short and longer term PLM use with patient characteristics

SECONDARY OUTCOMES:
Rate of Usability of PLM | 6 Months
  Usability (how useful they found PLM, what parts of the site they used, etc.) will be assessed using a patient experience survey at the end of the study
Rate of Overall Satisfaction with PLM | 6 Months
  Satisfaction with the PLM experience wil be assessed using a 'patient experience' survey at the end of the study
Rate of Desirability with PLM | 6 Months
  Desirability (how much they enjoyed using PLM, etc) wil be assessed using a patient experience survey at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Freedman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Occhiogrosso RH, Ren S, Tayob N, Li T, Gagnon HC, Paz A, Freedman RA. Feasibility of an Online Patient Community to Support Older Women With Newly Diagnosed Breast Cancer. Clin Breast Cancer. 2022 Feb;22(2):178-185. doi: 10.1016/j.clbc.2021.06.004. Epub 2021 Jun 12. PMID 34275766